CLINICAL TRIAL: NCT01833325
Title: A Pilot Study to Assess the Safety of Proton Therapy for Subfoveal Neovascularization Associated With Age-Related Macular Degeneration
Brief Title: Proton Radiation Therapy for Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UFPTI 1206-EY01
Record Dates: First submitted 2013-03-27; First posted 2013-04-16 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age-Related Macular Degeneration; Macular Degeneration; Proton radiation; Choroidal Neovascular Membranes
MeSH Terms: conditions — Macular Degeneration | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton radiation (Experimental): Proton radiation given to a total dose of 24 cobalt gray equivalent (CGE) in 2 treatments
  Interventions: Radiation: Proton radiation

INTERVENTIONS:
Radiation: Proton radiation — Proton radiation given to a total dose of 24 cobalt gray equivalent (CGE) in 2 treatments

SUMMARY:
This is a pilot study to determine if proton radiation therapy can provide effective and safe treatment for subfoveal neovascularization membrane (SNVM). The study will include adult patients over the age of 50 with macular degeneration, who have subfoveal neovascularization membrane (SNVM) and have had prior treatment with Avastin or Lucentis. Additional purposes of this study are to see if the growth of neovascular membranes can be stopped and overall vision improved with the use of protons and assess the side effects associated with this treatment.

DETAILED DESCRIPTION:
As part of this study, participants will have had a standard of care comprehensive eye exam by an Ophthalmologist to include visual acuity, fundus photography, fluorescein angiography and optical coherence tomography prior to treatment.

Participants will receive radiation using protons for 2 consecutive days. Each treatment will take 30 minutes. They will receive a total dose of 24 cobalt gray equivalent (CGE) in 2 treatments. A total of 10 participants will be enrolled on this study.

A comprehensive eye exam by an Ophthalmologist will be performed 30 days after radiation treatment with protons. Additionally, a physical examination per a Radiation Oncologist including a toxicity evaluation and comprehensive eye exam by an Ophthalmologist will be performed every 3 months for 1 year following radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with subfoveal neovascular membranes identified on fluorescein angiography.
* Visual acuity (best corrected vision) 20/200 or worse in affected eye.
* Patient must be 50 years of age or older at time of consent.
* Patients must have had prior treatment for macular degeneration with Avastin (bevacizumab) or Lucentis (ranibizumab).
* Women must be post menopausal or have had a hysterectomy.

Exclusion Criteria:

* History of diabetes.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-05; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with acute and late morbidity of the eye as a measure of safety | 1 year after completion of radiation treatment
Number of participants with cessation of growth of neovascular membranes. | 1 year after completion of radiation treatment
Visual acuity per comprehensive eye exam | 1 year after completion of radiation treatment
Frequency of intravitreal injections following radiation treatment | 1 year after completion of radiation treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roi Dagan, MD,, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

REFERENCES:
- [Background] Macular Degeneration Foundation Adult Macular Degeneration. Available at: http://www.eyesight.org/Macular_Degeneration/Adult_MD/adult_md.html. Accessed March 8, 2012.
- [Background] Argon laser photocoagulation for senile macular degeneration. Results of a randomized clinical trial. Arch Ophthalmol. 1982 Jun;100(6):912-8. doi: 10.1001/archopht.1982.01030030920003. PMID 7046707
- [Background] Krypton laser photocoagulation for neovascular lesions of age-related macular degeneration. Results of a randomized clinical trial. Macular Photocoagulation Study Group. Arch Ophthalmol. 1990 Jun;108(6):816-24. doi: 10.1001/archopht.1990.01070080058036. PMID 1693496
- [Background] Bressler NM; Treatment of Age-Related Macular Degeneration with Photodynamic Therapy (TAP) Study Group. Photodynamic therapy of subfoveal choroidal neovascularization in age-related macular degeneration with verteporfin: two-year results of 2 randomized clinical trials-tap report 2. Arch Ophthalmol. 2001 Feb;119(2):198-207. PMID 11176980
- [Background] Laser photocoagulation of subfoveal neovascular lesions in age-related macular degeneration. Results of a randomized clinical trial. Macular Photocoagulation Study Group. Arch Ophthalmol. 1991 Sep;109(9):1220-31. doi: 10.1001/archopht.1991.01080090044025. PMID 1718250
- [Background] Chakravarthy U, Gardiner TA, Archer DB, Maguire CJ. A light microscopic and autoradiographic study of non-irradiated and irradiated ocular wounds. Curr Eye Res. 1989 Apr;8(4):337-48. doi: 10.3109/02713688908996381. PMID 2721224
- [Background] Plowman PN, Harnett AN. Radiotherapy in benign orbital disease. I: Complicated ocular angiomas. Br J Ophthalmol. 1988 Apr;72(4):286-8. doi: 10.1136/bjo.72.4.286. PMID 3378026
- [Background] Macfaul PA, Bedford MA. Ocular complications after therapeutic irradiation. Br J Ophthalmol. 1970 Apr;54(4):237-47. doi: 10.1136/bjo.54.4.237. No abstract available. PMID 5310660
- [Background] Guyer DR, Mukai S, Egan KM, Seddon JM, Walsh SM, Gragoudas ES. Radiation maculopathy after proton beam irradiation for choroidal melanoma. Ophthalmology. 1992 Aug;99(8):1278-85. doi: 10.1016/s0161-6420(92)31832-9. PMID 1325044
- [Background] Chakravarthy U, Houston RF, Archer DB. Treatment of age-related subfoveal neovascular membranes by teletherapy: a pilot study. Br J Ophthalmol. 1993 May;77(5):265-73. doi: 10.1136/bjo.77.5.265. PMID 8318462
- [Background] Yonemoto LT, Slater JD, Blacharski P, Archambeau JO, Loredo LN, Oeinck SC, Teichman S, Moyers M, Slater JM. Dose Response in the Treatment of Subfoveal Choroidal Neovascularization in Age-Related Macular Degeneration: Results of a Phase I/II Dose-Escalation Study Using Proton Radiotherapy. Journal of Radiosurgery. 2000;3(1):47-54. DOI: 10.1023/A:1009525220716
- [Background] Zambarakji HJ, Lane AM, Ezra E, Gauthier D, Goitein M, Adams JA, Munzenrider JE, Miller JW, Gragoudas ES. Proton beam irradiation for neovascular age-related macular degeneration. Ophthalmology. 2006 Nov;113(11):2012-9. doi: 10.1016/j.ophtha.2006.05.036. Epub 2006 Aug 28. PMID 16935343
- [Background] Brown DM, Kaiser PK, Michels M, Soubrane G, Heier JS, Kim RY, Sy JP, Schneider S; ANCHOR Study Group. Ranibizumab versus verteporfin for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1432-44. doi: 10.1056/NEJMoa062655. PMID 17021319
- [Background] Sivagnanavel V, Evans JR, Ockrim Z, Chong V. Radiotherapy for neovascular age-related macular degeneration. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD004004. doi: 10.1002/14651858.CD004004.pub2. PMID 15495075
- [Background] Park SS, Daftari I, Phillips T, Morse LS. Three-year follow-up of a pilot study of ranibizumab combined with proton beam irradiation as treatment for exudative age-related macular degeneration. Retina. 2012 May;32(5):956-66. doi: 10.1097/IAE.0b013e31822a8d6a. PMID 22183743
- [Derived] Evans JR, Igwe C, Jackson TL, Chong V. Radiotherapy for neovascular age-related macular degeneration. Cochrane Database Syst Rev. 2020 Aug 26;8(8):CD004004. doi: 10.1002/14651858.CD004004.pub4. PMID 32844399